CLINICAL TRIAL: NCT00316238
Title: A Double-Blind Dose-Response Study Comparing Rapid Acting Intramuscular Olanzapine and Intramuscular Placebo in Agitated Patients With Schizophrenia
Brief Title: A Study Using Rapid Acting Intramuscular Olanzapine in Agitated Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5294; F1D-JE-RA02
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: olanzapine-RAIM
Drug: placebo

SUMMARY:
To investigate dose-response of Rapid Acting Intramuscular Olanzapine in Agitated Patients with Schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia that meets disease diagnostic criteria in DSM-IV-TR
* Patients must be inpatients during the study
* Patients must have a minimum total score of no less than 14 on the five items of the PANSS-EC and at least one individual item score of no less than 4 using the 1-7 scoring system prior to the first injection of study drug

Exclusion Criteria:

* Patients who have a known history of diabetes mellitus.
* Patients who have received treatment with antipsychotics or other prohibited concomitant medicines within 2 hours prior to the first IM study drug administration
* Patients who have had treatment with benzodiazepines within 4 hours prior to first IM study drug administration.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate dose-response relationship and to confirm the efficacy of IM olanzapine by sequentially comparing each of IM olanzapine groups and IM placebo group with respect to the changes from baseline to 2 hours post first IM injection of agitation.

SECONDARY OUTCOMES:
To determine if the efficacy of IM olanzapine is greater than IM placebo by evaluating sequentially comparing changes at 30 min, 60 min, 90 min post first IM injection of agitation, as measured by the PANSS-EC in schizophrenia patients.
To determine if the efficacy of IM olanzapine groups are greater than the IM placebo by evaluating sequentially changes from baseline to 2 hours post first IM injection in the rate of responder, CGI-I, and ACES.
To examine whether a dose-response relationship exists for IM olanzapine in higher agitation, by using mean changes of PANSS-EC total score from baseline to 2 hours post first IM injection as measured by PANSS-EC (Score total no less than 20).
To compare the efficacy of IM olanzapine(2.5, 5, 7.5, or 10 mg) to IM placebo by evaluating sequentially changes from baseline to 24 hours post first IM injection in the PANSS-EC, CGI-S, Clinical Global Impression-Improvement of Illness (CGI-), and ACES.
To compare efficacy of IM olanzapine(2.5, 5, 7.5, or 10 mg)to IM placebo in the frequency of patients who need second injection and time to second injection.
To compare the safety of IM olanzapine groups to IM placebo group over a 24 hours period in terms of ACES, TEAE, changes in laboratory values, pulse, blood pressure, ECG, DIEPSS.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Japan (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tottori
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamagata

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com